CLINICAL TRIAL: NCT03235076
Title: Investigation of Pharmacokinetics, Safety, Tolerability and Pharmacodynamic Effects of a Single Oral 10 mg BAY1101042 MR Tablet Dose in Male and Female Subjects With Renal Impairment and in Age-, Gender-, and Weight- Matched Healthy Subjects in a Single Center, Non-controlled, Open-label, Observational Design
Brief Title: Clinical Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Pharmacodynamic Effects of a Single Oral 10 mg BAY1101042 Tablet Dose in Men and Woman With Renal Impairment and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18745; 2017-001141-28 (EudraCT Number)
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subjects with mild renal impairment (Experimental): Single oral dose of 10 mg BAY1101042 (given as 5 mg MR tablets)
  Interventions: Drug: BAY1101042
- Subjects with moderate renal impairment (Experimental): Single oral dose of 10 mg BAY1101042 (given as 5 mg MR tablets)
  Interventions: Drug: BAY1101042
- Subjects with severe renal impairment (Experimental): Single oral dose of 10 mg BAY1101042 (given as 5 mg MR tablets)
  Interventions: Drug: BAY1101042
- Matched healthy subject group (Experimental): Single oral dose of 10 mg BAY1101042 (given as 5 mg MR tablets)
  Interventions: Drug: BAY1101042

INTERVENTIONS:
Drug: BAY1101042 — Single oral dose of 10 mg BAY 1101042 (given as 5 mg MR tablets)

SUMMARY:
To investigate the pharmacokinetics of BAY1101042 in subjects with mild to severe renal impairment, stratified according to estimated glomerular filtration rate (eGFR) determined 2-10 days prior to dosing, and age-, weight- and gender- matched healthy subjects and to assess the safety, tolerability, and pharmacodynamics of BAY1101042 after a single oral dose of a 10 mg BAY1101042 given as 5 mg modified release (MR) tablet.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and follow study-related instructions and ability to participate in the study for the entire period.
* Age: 18 to 79 years (inclusive) at the screening visit.
* Body mass index (BMI): 18 to 34 kg/m² (both inclusive).
* Male or female subject.
* Only women without childbearing potential will be included in the study (e.g. postmenopausal for at least one year, women with bilateral ovariectomy and women with hysterectomy).

Subjects with renal impairment:

* eGFR <90 mL/min/1.73 m*2 determined from serum creatinine 2-10 days prior to dosing.
* Stable renal disease, i.e. a serum creatinine value determined at least 3 months before the pre-study visit (e.g. during routine diagnostics) should not vary by more than 20% from the serum creatinine value determined at the pre-study visit.

Healthy subjects:

- eGFR ≥90 mL/min/1.73 m*2 determined from serum creatinine 2-10 days prior to dosing.

Exclusion Criteria:

* Pregnant or lactating women.
* Medical disorder, condition or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve from zero to infinity after single dose (AUC) of BAY1101042 | Study Day 1 to Study Day 6
  Area under the concentration vs. time curve from zero to infinity after single dose of BAY1101042
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of BAY1101042 | Study Day 1 to Study Day 6
  Maximum observed concentration of BAY1101042 in plasma after single dose administration
AUCu of BAY1101042 | Study Day 1 to Study Day 6
  Area under the unbound concentration vs. time curve from zero to infinity after single dose of BAY1101042
Cmax,u of BAY1101042 | Study Day 1 to Study Day 6
  Maximum observed unbound concentration of BAY1101042 in plasma after single dose administration of BAY1101042

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany